CLINICAL TRIAL: NCT07175415
Title: ITCC-104: HEM-iSMART International Proof of Concept Therapeutic Stratification Trial of Molecular Anomalies in Relapsed or Refractory HEMatological Malignancies in Children, Sub-Protocol E: Capivasertib + Venetoclax + Dexamethasone in Pediatric Patients With Relapsed or Refractory Hematological Malignancies
Brief Title: HEM-iSMART E: Capivasertib + Venetoclax + Dexamethasone in Pediatric Patients With Relapsed or Refractory Hematological Malignancies
Acronym: HEM-iSMART E
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: AstraZeneca (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-523132-39-00
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma (Precursor B-Lymphoblastic Lymphoma/Leukaemia) Recurrent; Lymphoblastic Lymphoma (Precursor B-Lymphoblastic Lymphoma/Leukaemia) Refractory; Lymphoblastic Lymphoma (Precursor T-Lymphoblastic Lymphoma/Leukaemia) Recurrent; Lymphoblastic Lymphoma (Precursor T-Lymphoblastic Lymphoma/Leukaemia) Refractory
Keywords: Acute lymphoblastic leukemia; relapse; biomarker driven clinical trial; refractory; capivasertib; venetoclax; children; adolescents; young adults; lymphoblastic lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — capivasertib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capivasertib + Venetoclax + Dexamethasone (Experimental): Sub-study E: Each cycle lasts 28 days. Cycle 1: All patients in cycle 1 will receive 4 blocks of of capivasertib (days D4-7, 11-14, 18-21, 25-28), 28 days of venetoclax (days 1-28), and one block of seven days of dexamethasone (days 1-7). A 1-day venetoclax ramp-up is proposed in this study. Cycle 2 and subsequent cycles: similar to cycle 1. Patients in dose level -1, receive a lower dose of venetoclax. Patients in dose level 2 receive a higher dose of capivasertib. All patients receive age adapted intrathecal chemotherapy.
  Interventions: Drug: Capivasertib; Drug: Venetoclax; Device: Dexamethasone; Drug: Intrathecal chemotherapy

INTERVENTIONS:
Drug: Capivasertib — Oral
Drug: Venetoclax — Oral
Device: Dexamethasone — oral/intravenous
Drug: Intrathecal chemotherapy — IT: Methotrexate +/- prednisone/hydrocortisone/cytarabine according to the degree of central nervous involvement

SUMMARY:
HEM-iSMART is a master protocol which investigates multiple investigational medicinal products in children, adolescents and young adults (AYA) with relapsed/refractory (R/R) ALL and LBL. Sub-protocol E is a phase I/II trial evaluating the safety and efficacy of capivasertib + venetocolax in combination with dexamethasone in children and AYA with R/R ped ALL/LBL whose tumor present with alterations of the PAM pathway, or lacking any mutations.

DETAILED DESCRIPTION:
HEM-iSMART is a master protocol with sub-protocols. The overarching objective is that introducing targeted therapy using a biomarker driven approach for treatment stratification may improve the outcome of children with R/R acute lymphoblastic leukemia (ALL) and lymphoblastic lymphoma (LBL) It is characterized by a shared framework that allows for the investigation of multiple IMPs and generate pivotal safety and efficacy evidence within the sub-protocols to establish and define the benefits and risks of new treatments for children with R/R leukemia.

Sub-protocol E within HEM-iSMART is a phase I/II, multicenter, international, open-label clinical trial designed to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of capivasertib + venetoclax in combination with dexamethasone in children, adolescents and young adults with relapsed or refractory (R/R) hematological malignancies including ALL and LBL. Patients in must present alterations of the PAM pathway, or can be enrolled on a generic base lacking any mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Children ≥ 2 years and ≤ 18 years of age at the time of first diagnosis and less than 21 years at the time of inclusion
2. Performance status: Karnofsky performance status (for patients >16 years of age) or Lansky Play score (for patients ≤16 years of age) ≥ 50% (Appendix I).
3. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study specific screening procedures are conducted, according to local, regional or national guidelines.
4. For all oral medications patients must be able to comfortably swallow tablets (except for those for which the AAF is available; nasogastric or gastrostomy feeding tube administration is allowed only if indicated).
5. Patients must have had advanced molecular profiling and flow-cytometric analysis of their recurrent or refractory disease at a time-point before the first inclusion into this trial (see section 9.1 of the master protocol for detailed description of the molecular diagnostics required). Drug response profiling and methylation is highly recommended but not mandatory. Patients with advanced molecular profiling at diagnosis may be allowed to be included after discussion with the sponsor.
6. In the Phase II portion of the trial, 30% of the eligible patients will have to show alterations in the PI3K/AKT/mTOR pathway as follows: PI3K (including PIK3CA, PIK3CB, PIK3R1), AKT and loss of PTEN.
7. Patients with spinal cord compression should be deemed clinically stable prior to enrolment into the trial.
8. Adequate organ function:

RENAL AND HEPATIC FUNCTION (Assessed within 48 hours prior to C1D1):

* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) for age or calculated creatinine clearance as per the Schwartz formula or radioisotope glomerular filtration rate ≥ 60 mL/min/1.73 m2.
* Direct bilirubin ≤ 2 x ULN (≤ 3.0 × ULN for patients with Gilbert's syndrome).
* Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 5 x ULN; aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT ≤ 5 x ULN.

CARDIAC FUNCTION:

* Shortening fraction (SF) >29% (>35% for children < 3 years) and/or left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography.
* Absence of mean resting QTcF prolongation obtained from triplicate ECG performed at screening according to age group: (aged <12 years of age QTcF >440msec) (aged ≥12 years QTcF >450msec), using the Fridericia correction [QTcF formula]) or other clinically significant ventricular or atrial arrhythmia.

Exclusion Criteria:

1. Pregnancy or positive pregnancy test (urine or serum) in females of childbearing potential. Pregnancy test must be performed within 7 days prior to C1D1.
2. Sexually active participants of childbearing potential not willing to use highly effective contraceptive method (pearl index <1) as defined in CTFG HMA 2020 (Appendix II) during trial participation and until 30 days after end of study intervention for females and 16 weeks for males.
3. Breast feeding.
4. History of another primary malignancy.
5. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome) in case of oral IMPs.
6. Patients whose tumor present known mutations conferring resistance to venetoclax (e.g. BCL2 mutations of venetoclax binding-site (Gly101Val mutation, Phe104Leu/Cys mutations) and capivasertib (e.g. mutations in TSC1, TSC2 and STK11).
7. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to the study drugs, or drugs chemically related to study treatment or excipients that contraindicate their participation, including corticoids.
8. Known active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
9. Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion.
10. Subjects unwilling or unable to comply with the study procedures.
11. Previous treatment with capivasertib and venetoclax in combination (Patients who have previously received venetoclax in alternative combinations can be eligible for this sub-protocol. Patients previously treated with capivasertib are not eligible).
12. Current use of a prohibited medication or herbal preparation or requires any of these medications during the study. See Section 7, Appendix III for details. In general, strong and moderate inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort). In addition, participants should avoid herbal supplements and ingestion of large amounts of foods and beverages known to potently modulate CYP3A4 enzyme activity during study treatment.
13. Drugs known to significantly prolong the QT interval and associated with torsade de points (TdP) within 5 half-lives of the first dose of study treatment. Clinically significant electrolyte abnormalities associated with QTc prolongation and/or any factors, that in the judgement of the investigator may significantly increase the risk of QTc prolongation. History of QTc prolongation, congenital long QT syndrome, medical history significant for arrhythmia which is not resolved.
14. Patients who have consumed grapefruit, grapefruit products, Seville oranges (Including marmalade containing Seville oranges) or starfruit within 72 hours prior to the first dose of study drug.
15. Unresolved toxicity greater than NCI CTCAE v 5.0 ≥ grade 2 from previous anti-cancer therapy, including major surgery, except those that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profile of the study treatment (e.g., alopecia and/or peripheral neuropathy related to platinum or vinca alkaloid based chemotherapy) (Common Terminology Criteria for Adverse Events (CTCAE) (cancer.gov).
16. Active acute graft versus host disease (GvHD) of any grade or chronic GvHD of grade 2 or higher. Patients receiving any agent to treat or prevent GvHD post bone marrow transplant are not eligible for this trial.
17. Received immunosuppression post allogenic HSCT within one month of study entry.
18. Metabolic disorders:

    o HbA1c ≥8.0% (63.9 mmol/mol)
19. Wash-out periods of prior medication:

    1. CHEMOTHERAPY: At least 7 days must have elapsed since the completion of cytotoxic therapy, with the exception of hydroxyurea, 6-mercaptopurine, oral methotrexate and steroids which are permitted up until 48 hours prior to initiating protocol therapy. Patients may have received intrathecal therapy (IT) at any time prior to study entry.
    2. RADIOTHERAPY: Radiotherapy (non-palliative) within 21 days prior to the first dose of drug.
    3. HEMATOPOIETIC STEM CELL TRANSPLANTATION (HSCT):

       * Autologous HSCT within 2 months prior to the first study drug dose.
       * Allogeneic HSCT within 3 months prior to the first study drug dose.
    4. IMMUNOTHERAPY: At least 42 days must have elapsed after the completion of any type of immunotherapy, including CAR-T cell therapy other than monoclonal antibodies (e.g. Inotuzumab)
    5. MONOCLONAL ANTIBODIES AND INVESTIGATIONAL DRUGS: At least 21 days or 5 times the half-life (whichever is shorter) from prior treatment with monoclonal antibodies or any investigational drug under investigation must have elapsed before the first study drug.
    6. SURGERY: Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2031-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) / Recommended phase 2 dose (RP2D). | 2 years
  Defined as the highest dose level tested at which 0/6 or 1/6 patients experiences dose limiting toxicities (DLT) during course 1 with at least 2 patients experiencing DLT at the next higher dose.
Phase II: Best Overall Response Rate (ORR). | 4 years
  For patients with leukemia: CR and MRD response after 1 cycle of treatment. This includes determination of CR, CRp, CRi and minimal residual disease (MRD) negativity rate in patients suffering from overt morphological relapse of T-ALL at time of enrolment (morphological disease (M2/M3)), and the MRD negativity rate in those that entered with high-MRD levels but in morphological CR. These results will together be presented as a composite endpoint Overall Response rate (ORR). MRD negativity will be defined as ≤1x10-4 as generated by multi-parameter flow cytometry. For patients with lymphoma: Response in LBL patients is defined as CR, PR, minor response (MR) as defined in International pediatric NHL response criteria. In case of bone-marrow involvement MRD will be taken into account. For patients with lymphoma: Response in LBL patients is defined as CR, PR, minor response (MR) as defined in International pediatric NHL response criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Defined as time from C1D1 until death of any cause.
Event-free survival (EFS) | 5 years
  Defined as time from C1D1 to the first event (subsequent relapse after CR (including molecular reappearance), death of any cause, failure to achieve remission (CR, CRp or CRi), or secondary malignancy).
Cumulative incidence of relapse (CIR) | 5 years
  Estimate of the risk, that a patient will develop a relapse over a specified period of time.
Number of patients proceeding to hematopoietic stem cell transplantation (HSCT) after the experimental therapy. | 5 years
  The rate of those proceeding to subsequent allogenic HSC
Cumulative overall response rate (ORR) | 5 years
  Defined as the CR, CRp, CRi and MRD negativity rates after more than 1 cycle of treatment.
Rate of dose limiting toxicities (DLTs) | 5 years
  Number of participants with dose limiting toxicities (DLTs)
Peak Plasma Concentration (Cmax) | 4 years
  Estimation of venetoclax and dasatinib Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Lissat, MD PhD, Principal Investigator — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No